CLINICAL TRIAL: NCT01861509
Title: Pharmacokinetic, Pharmacodynamic and Interleukin Profile of Intramuscularly Administered BP-C1 in Women With Metastatic Breast Cancer. A Phase ID Study
Brief Title: BP-C1 in Metastatic Breast Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Meabco A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BMC2012-4
Record Dates: First submitted 2013-05-13; First posted 2013-05-23 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Metastatic Breast Cancer; Stage IV Breast Cancer
Keywords: BP-C1; Metronomic chemotherapy; Platinum analogue; Cis-diammineplatinum(II) complexed with a polymer containing benzene polycarboxylic acids derived from lignin; Benzene polycarboxylic acids complex with cis-diammineplatinum(II); Breast cancer; Cisplatin; Metastatic Breast Cancer; Cis-diammineplatinum(II) complex, containing mono-deprotonated benzene-poly-carboxylic acids, derived from lignin, and hydroxyl group as O-donor ligands
MeSH Terms: conditions — Breast Neoplasms | interventions — Hydroxyl Radical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BP-C1 IM Injections (Experimental): BP-C1 given in daily intramuscular doses of 0.035 mg/kg bodyweight in one syringe per day during a total treatment of 32 days.
  Interventions: Drug: BP-C1

INTERVENTIONS:
Drug: BP-C1 — BP-C1, 0.05% solution for injection; doses: 0.035 mg/kg body weight (0.07 mL/kg) intramuscularly once daily for 32 consecutive days
  Other Names: Cis-diammineplatinum(II) complexed with a polymer containing benzene polycarboxylic acids derived from lignin; Benzene polycarboxylic acids complex with cis-diammineplatinum(II); Cis-diammineplatinum(II) complex, containing mono-deprotonated benzene-poly-carboxylic acids, derived from lignin, and hydroxyl group as O-donor ligands

SUMMARY:
This study is an open label, non-randomized phase I single-armed study in women with metastatic breast cancer (MBC) who have previously undergone all available standard chemotherapy regimens. The purpose of the study is to estimate the pharmacokinetics (PK) after single dose and multiple dose of BP-C1, investigate interleukin levels during BP-C1 treatment and assess treatment response according to RECIST criteria.

DETAILED DESCRIPTION:
BP-C1, solution for injections 0.05%, is currently being developed for treatment of patients with metastatic breast cancer with palliative intent.

Active substance of the product, which is a novel platinum-containing anticancer agent developed for intramuscular administration, is а cis-diammineplatinum(II) complexed with a polymer containing benzene polycarboxylic acids derived from lignin.

The amphiphilic characteristics of the polymer have resulted in a product with clear and significantly altered and improved properties compared to other platinum analogues, e.g. cisplatin, carboplatin and oxaliplatin.

BP-C1 preserves antitumour activity of its predecessors (e.g. cisplatin and carboplatin), additionally offering the following advantages that ensure favourable outcome of treatment of metastatic breast cancer patients:

* injectable solution (intramuscular) does not cause injection site reactions;
* can be administered at home by a nurse or a patient;
* has an improved pharmacokinetic profile;
* demonstrates efficacy comparable to cisplatin and much higher than carboplatin (in-vitro; in-vivo data);
* exerts an additional immunomodulatory activity.

In this study six female patients with MBC who have previously undergone at least third line therapy will be enrolled. Each included patient will participate in a screening period (maximum duration of 21 days) following by 32-day treatment period and 28-day follow-up period.

The patients will be treated with BP-C1(daily intramuscular injections) for 32 consecutive days. The study is undertaken to evaluate pharmacokinetics, pharmacodynamics and treatment effect of BP-C1.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with metastatic breast cancer (MBC, stage IV).
2. 18 and 80 years of age.
3. Measurable lesions / lymph nodes.
4. Have previously undergone at least third line chemotherapy.
5. Expected survival time at least 3 months.

Exclusion Criteria:

1. Abnormal liver function classified as total bilirubin >34 μmol/L or ALAT > 3 times the upper limit of normal range (ULN). In case of metastases in the liver, the ALAT limit for exclusion is set to 5xULN. Re-test results of blood samples taken again up to 2 days before Day-1 must keep meeting eligibility criteria.
2. Abnormal kidney function defined by serum creatinine >120 μmol/L. Re-test results of blood samples taken again up to 2 days before Day-1 must keep meeting eligibility criteria.
3. Abnormal coagulation capacity defined by the relative arbitrary concentration of coagulation factors 2,7,10 INR >1.3. Re-test results of blood samples taken again up to 2 days before Day-1 must keep meeting eligibility criteria.
4. Brain metastases in symptomatic patients requiring ≥4 mg dexamethasone/day. However, patients with treated brain metastases by surgery or radiation who are stable and symptom-free (<4 mg dexamethasone/day) for a minimum period of 4 weeks prior to study treatment are eligible.
5. Synchronous cancer except for non-melanoma skin cancer and early stage of cervical cancer.
6. Abnormal haematology status defined by Hb < 9.0 g/dL, platelet count < 75,000/mm^3 and leukocytes < 3x10^9/L. Re-test results of blood samples taken again up to 2 days before Day-1 must keep meeting eligibility criteria.
7. Clinically significant abnormal ECG.
8. Karnofsky Performance Status Score < 50%.
9. Pregnant or breast feeding women.
10. Women of fertile age who do not want to be tested for possible pregnancy.
11. Fertile female who do not want to use safe protection against pregnancy, starting one month before start of the trial treatment and lasting at least six weeks after.
12. Uncontrolled bacterial, viral, fungal or parasite infection.
13. Under systemic treatment with corticosteroids or other immunosuppressive drugs during the last 21 days before start of the trial treatment. Systemic treatment with <4 mg dexamethasone/day is allowed
14. Participating in another clinical trial with pharmaceuticals during the last six weeks before start of this trial treatment.
15. Not able to understand written or oral information.
16. Do not want or is not able to give written consent to participate in the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01-19 (Actual); Primary Completion 2016-01-20 (Actual); Study Completion 2016-01-20 (Actual)

PRIMARY OUTCOMES:
Single-dose PK: Maximum Observed Serum Concentration (Cmax) for Platinum | Pre-dose, 10, 20, 30, 35, 40, 45, 60, 120 min and 6, 24, 48 hours post dose
  Maximum Observed Serum Concentration (Cmax) for Platinum after the single dose of BP-C1 during the period of Day-1 to Day 1
Single-dose PK: Time to Reach Maximum Observed Serum Concentration (Tmax) for Platinum | Pre-dose, 10, 20, 30, 35, 40, 45, 60, 120 min and 6, 24, 48 hours post dose
  Time to Reach Maximum Observed Serum Concentration (Tmax) for Platinum after the single dose of BP-C1 during the period of Day-1 to Day 1
Single-dose PK: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUC(0-t)) for Platinum | Pre-dose, 10, 20, 30, 35, 40, 45, 60, 120 min and 6, 24, 48 hours post dose
  AUC(0-t) = Area under the serum concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration after the single dose of BP-C1 during the period of Day-1 to Day 1
Single-dose PK: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC(0-∞)) | Pre-dose, 10, 20, 30, 35, 40, 45, 60, 120 min and 6, 24, 48 hours post dose
  after the single dose of BP-C1 during the period of Day-1 to Day 1
Single-dose PK: Serum Decay Half-Life (T1/2) for Platinum | Pre-dose, 10, 20, 30, 35, 40, 45, 60, 120 min and 6, 24, 48 hours post dose during the period of Day-1 to Day 1
  Serum decay half-life is the time measured for the serum concentration of Platinum to decrease by one half after the single dose of BP-C1 during the period of Day-1 to Day 1
Multiple-dose PK: Maximum Observed Serum Concentration at Steady State (Css,max) for Platinum | Pre-dose, 10, 20, 30, 35, 40, 45, 60, 120 min and 6, 24, 48 hours post dose
  Maximum Observed Serum Concentration at steady state (Css,max) for Platinum during the period of Day 32 to Day 34
Multiple-dose PK: Time to Reach Maximum Observed Serum Concentration at steady state (Tss,max) for Platinum | Pre-dose, 10, 20, 30, 35, 40, 45, 60, 120 min and 6, 24, 48 hours post dose
  Time for Css,max at steady state for Platinum during the period of Day 32 to Day 34
Multiple-dose PK: Minimum Observed Serum Concentration at Steady State (Css,min) for Platinum | Pre-dose, 10, 20, 30, 35, 40, 45, 60, 120 min and 6, 24, 48 hours post dose
  Minimum Observed Serum Concentration at Steady State (Css,min) for Platinum during the period of Day 32 to Day 34
Multiple-dose PK: Average Serum concentration at steady state (Css,av) for Platinum | Pre-dose, 10, 20, 30, 35, 40, 45, 60, 120 min and 6, 24, 48 hours post dose
  Average Serum concentration at steady state (Css,av) for Platinum during the period of Day 32 to Day 34
Multiple-dose PK: Area Under the Curve within a dosing interval of tau (=24 hr) at steady state (AUCss,tau) for Platinum | Pre-dose, 10, 20, 30, 35, 40, 45, 60, 120 min and 6, 24, 48 hours post dose
  Area under the serum concentration versus time curve within a dosing interval of tau (=24 hr) at steady state (AUCss,tau) during the period of Day 32 to Day 34
Multiple-dose PK: Serum Decay Half-Life (T1/2) for Platinum | Pre-dose, 10, 20, 30, 35, 40, 45, 60, 120 min and 6, 24, 48 hours post dose
  Serum decay half-life is the time measured for the plasma concentration of Platinum to decrease by one half during the period of Day 32 to Day 34

SECONDARY OUTCOMES:
Interleukin Serum levels (Interferon γ and β, Tumour Necrosis Factor (TNF-α), IL-1beta, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12, IL-21 and IL-25) | Day-1, Day 1, Day 16, Day 32, Day 34
Change (%) in the sum of diameters of target lesions | baseline to Day 32 of treatment
  Diameter of target lesions will be measured by computer tomography (CT) with contrasting using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Number of target lesions | baseline to Day 32 of treatment
  Number of target lesions per each patient will be evaluated by CT with contrasting. Change in number of target lesions from baseline to Day 32 of treatment will be presented in shift tables
Treatment response | baseline to Day 32 of treatment
  In accordance with RECIST v1.1 the treatment response will be classified as 'complete response', 'partial response', 'stable disease' or 'progressive disease': Complete response (CR): disappearance of all target lesions. Partial response (PR): at least 30% decrease in the sum of longest diameters of target lesions, taking as reference the baseline sum of diameters. Progressive disease (PD): at least 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum might also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions will also be considered progression. Stable disease (SD): neither sufficient shrinkage to qualify for PR, nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study

CONTACTS AND LOCATIONS:
Overall Officials: Stig Larsen, Prof., Study Director — Meabco A/S
Locations (2):
- Oncology Unit. Sheba Medical Centre, Ramat Gan, Israel
- Lampang Cancer Center, Lampang, Thailand

IPD SHARING:
Plan to Share IPD: No